CLINICAL TRIAL: NCT00045500
Title: A Phase I Trial Of UCN-01 And Prednisone In Patients With Refractory Solid Tumors And Lymphomas
Brief Title: UCN-01 and Prednisone in Treating Patients With Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000256599; NCI-02-C-0241; NCI-5694; NCT00041873 (obsolete NCT alias)
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2005-08

CONDITIONS: Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; intraocular lymphoma; primary central nervous system non-Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult T-cell leukemia/lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent mantle cell lymphoma; unspecified adult solid tumor, protocol specific; recurrent adult Burkitt lymphoma; recurrent grade 3 follicular lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Hodgkin Disease; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Burkitt Lymphoma; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — 7-hydroxystaurosporine; Prednisone

INTERVENTIONS:
Drug: 7-hydroxystaurosporine
Drug: prednisone

SUMMARY:
RATIONALE: UCN-01 may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining UCN-01 with prednisone may kill more cancer cells.

PURPOSE: Phase I trial to study the effectiveness of combining UCN-01 with prednisone in treating patients who have refractory solid tumors or lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of UCN-01 in combination with prednisone in patients with refractory solid tumors or lymphomas.
* Determine the toxic effects of this regimen in these patients.
* Assess the pharmacokinetics of this regimen in these patients.
* Assess any tumor response in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of UCN-01.

Patients receive oral prednisone daily on days 1-5 and UCN-01 IV over 36-72 hours on days 3-5. Courses repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of UCN-01 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the recommended phase II dose.

Patients are followed every 3-12 months for 5 years.

PROJECTED ACCRUAL: Approximately 24 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor or lymphoma

  * Progressive disease after standard therapy
  * No other therapy is likely to improve survival
* Prostate cancer patients must have progressed through hormonal therapy with gonadotropin-releasing hormone (GnRH) agonists and withdrawal of testosterone receptor antagonists

  * Patients must continue on GnRH agonist during study (if orchiectomy has not been performed) and have castrate testosterone levels
* Brain metastases allowed if treated and the patient has been stable off anti-seizure medication or steroids for > 6 months
* No local complications from disease requiring urgent therapy (i.e., hydronephrosis, spinal cord compression, or severe pain requiring improved pain management)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count greater than 1,000/mm^3
* Platelet count greater than 100,000/mm^3
* 12-hour fasting glucose no greater than 110 mg/dL OR
* 12-hour fasting glucose no greater than 140 mg/dL with hemoglobin A1C no greater than 6.5 mg/dL

Hepatic

* PT/PTT no greater than 1.5 times upper limit of normal (ULN)
* Bilirubin no greater than 1.5 times ULN (unless Gilbert's syndrome present)
* AST/ALT no greater than 2.5 times ULN

Renal

* Creatinine clearance greater than 60 mL/min OR
* Creatinine no greater than 1.5 mg/dL

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris

Pulmonary

* No interstitial lung disease within the past year
* No requirement for oxygen therapy for hypoxia in the past 6 months

Gastrointestinal

* No diagnosis of duodenal or gastric ulcer
* No severe gastritis within the past 6 months

Other

* HIV negative
* No prior allergic reactions to other indolocarbazoles
* No diabetes or hyperglycemia within the past year that required a diabetic diet, oral hypoglycemics, or insulin
* No other uncontrolled illness
* No active infection
* No seizure disorder
* No psychiatric illness that would preclude study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No prior UCN-01

Endocrine therapy

* See Disease Characteristics
* No other concurrent oral or IV steroids

Radiotherapy

* At least 4 weeks since prior radiotherapy and recovered

Surgery

* See Disease Characteristics
* At least 21 days since prior major surgery

Other

* See Disease Characteristics
* At least 4 weeks since prior investigational agents
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-06; Primary Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Melillo, MD, Study Chair — National Cancer Institute - Frederick
Locations (3):
- United States (3):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland
  - Frederick Cancer Research and Development Center, Frederick, Maryland